CLINICAL TRIAL: NCT05898841
Title: An Open Label, Comparative, Randomized , Phase IV Pilot Study to Evaluate the Efficacy and Safety of a Rilpivarine-based Antiretroviral Tratment Regimen in HIV- Infected Patients With Liver Metabolic Disease Who Maintain Udetectable HIV Viral Load
Brief Title: Study to Evaluate the Efficacy and Safety of a Rilpivarine-based Antiretroviral Tratment Regimen in HIV- Infected Patients With Liver Metabolic Disease Who Maintain Udetectable HIV Viral Load
Acronym: MAFALDA-R
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundacion SEIMC-GESIDA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GESIDA 12422
Record Dates: First submitted 2023-04-05; First posted 2023-06-12 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: HIV Infections; Fatty Liver Disease
MeSH Terms: conditions — HIV Infections; Non-alcoholic Fatty Liver Disease | interventions — dolutegravir; Rilpivirine; Tenofovir; tenofovir alafenamide; Emtricitabine; Racivir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dolutegravir (DTG) 50 mg/day + Rilpivirine (RPV) 25mg per day (Experimental): Dolutegravir (DTG) 50 mg/day + Rilpivirine (RPV) 25mg per day. They may be administered in combination as 50/25 mg/day tablets (Juluca 50/25) or separately as Dolutegravir 50 mg/d tablets together with Rilpivirine 25 mg/d tablets (Tivicay 50 + Edurant 25)
  Interventions: Drug: Dolutegravir (DTG) 50 mg/day + Rilpivirine (RPV) 25mg per day
- TDF 245 mg /day or TAF 25 mg /day + FTC 200 mg /day + RPV 25 mg / day (Experimental): Tenofovir disoproxil fumarate (TDF) 245 mg per day or Tenofovir alafenamide (TAF) 25 mg per day + Emtricitabina (FTC) 200 mg/d + Rilpivirina (RPV) 25 mg/d. They may be administered as single tablets (EVIPLERA 200 mg/25 mg/245 mg) or in combination forms where one tablet contains TDF/TAF and FTC and another RPV tablet (TDF/FTC + Edurant 25 or Descovy 25/200 + Edurant 25)
  Interventions: Drug: Tenofovir disoproxil fumarate (TDF) 245 mg per day or Tenofovir alafenamide (TAF) 25 mg per day + Emtricitabine (FTC) 200 mg per day + Rilpivirine 25 mg per day
- Continue with their previous treatment. Any previous HAART does not contain RILPIVIRINE. (Active Comparator): Patients who are randomised to this treatment arm will continue with the HAART they were receiving prior to signing the informed consent. As in arms 1 and 2, a change in the form of HAART administration (from a combined to a separate form and vice versa) will be allowed as long as the HAART components are respected.
  Interventions: Drug: Continue with their previous treatment. Any previous HAART that does not contain Rilpivirine.

INTERVENTIONS:
Drug: Dolutegravir (DTG) 50 mg/day + Rilpivirine (RPV) 25mg per day — DTG/RPV will be administered in combination as 50/25 mg/day tablets or separately as DTG 50 mg/d tablets together with RPV 25 mg/d tablets. There will be no problem if during the course of the study the patient is switched from the combined form to the separate form and vice versa as long as the HAART (Highly Active Antiretroviral Therapy) components are respected.
  Arms: Dolutegravir (DTG) 50 mg/day + Rilpivirine (RPV) 25mg per day
Drug: Tenofovir disoproxil fumarate (TDF) 245 mg per day or Tenofovir alafenamide (TAF) 25 mg per day + Emtricitabine (FTC) 200 mg per day + Rilpivirine 25 mg per day — TDF 245 mg/d or TAF 25mg/d together with FTC 200 mg/d and RPV 25 mg/d. They may be administered as single tablets or in combination forms where one tablet contains TDF/TAF and FTC and another RPV tablet. There will be no problem if during the course of the study the patient is switched from the combined form to the separate form and vice versa as long as the HAART components are respected.
  Arms: TDF 245 mg /day or TAF 25 mg /day + FTC 200 mg /day + RPV 25 mg / day
Drug: Continue with their previous treatment. Any previous HAART that does not contain Rilpivirine. — Patients who are randomised to this treatment arm will continue with the HAART they were receiving prior to signing the informed consent. As in arms 1 and 2, a change in the form of HAART administration (from a combined to a separate form and vice versa) will be allowed as long as the HAART components are respected.
  Arms: Continue with their previous treatment. Any previous HAART does not contain RILPIVIRINE.

SUMMARY:
In HIV-infected people with metabolic fatty liver disease and liver fibrosis of any degree, as measured by non-invasive testing, antiretroviral treatment that includes rilpivinire for 18 months results in a slowing of progression and/or reduction of fatty metabolic liver disease, attenuating inflammation and liver fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age with HIV infection who have never received antiretroviral treatment with Rilpivirine.
* Have a stable ART pattern for at least the last 6 month

Exclusion Criteria:

* Not having received more than three previous lines of antiretroviral treatment
* No resistance mutations that compromise the efficacy of Rilpivirine, Dolutegravir, Tenofovir (TDF and/or TAF) or Emtricitabine.
* Have an HIV viral load < 50 copies/ml for at least the last 6 months, 1 blip below 500 copies/ml is allowed during this period.
* Have an ultrasound-diagnosed fatty liver metabolic disease or a CAP (Controlled Attenuation Parameter®) measurement > 238 dB/m with an IQR < 30 dB/m.
* Have an fatty liver metabolic disease with some degree of fibrosis diagnosed by ET (Fibroscan®) > 5.2 kPa. In patients in whom ET is not possible, have a FIB-4 >1.3.
* Be able to understand and comply with the requirements and instructions of the protocol.
* Understanding long-term commitment to study
* Acceptance of their participation in the study by signing an informed consent form.

Exclusion Criteria:

* Have chronic HBV infection (presence of HBsAg+) or HCV (detectable HCV viral load). Patients with past treated HCV are also not allowed to be included (does not include patients with spontaneously resolved HCV infection).
* Have diabetes mellitus on treatment with SGLT2, GLP1 or plioglitazone of less than 6 months duration.
* Have a history of alcohol abuse
* Harmful alcohol consumption, defined as >30 grams of alcohol per day in men and >20 grams of alcohol per day in women.
* Have chronic decompensated liver disease, defined as any of the following: presence of encephalopathy, ascites, coagulopathy, oesophageal or gastric varices, or persistent jaundice.
* Any previous physical or mental condition (such as habitual drug use) that the investigator believes may interfere with the patient's ability to comply with the study protocol.
* Pregnancy or breastfeeding at the screening visit or at any time during the study or intention to become pregnant during the study period.
* Prior history of Rilpivirine use of any duration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2023-05-26 (Actual); Primary Completion 2025-07-07 (Actual); Study Completion 2025-07-07 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of Rilpivirine (RPV) as part of the antiretroviral treatment regimen in VIH-infected people, to slow the progression and/or reduce liver fibrosis of any degree | 18 months
  To measure the no progression and/or regression of liver fibrosis:
  No change in liver stiffness as measured by ET (Transient Elastography) or FIB4 at the 18-month visit with respect to the baseline, the intervention group (branches 1 and 2) compared to the control group.
To evaluate the efficacy of Rilpivirine (RPV) as part of the antiretroviral treatment regimen in VIH-infected people, to slow the progression and/or reduce liver fibrosis of any degree | 18 months
  Reduction in liver stiffness measured by ET or FIB4 at the 18-month visit from baseline in the intervention group (arms 1 and 2) versus the control group.

SECONDARY OUTCOMES:
Efficacy of RPV in reducing liver fibrosis of any grade | 12-18 months
  To evaluate the efficacy of RPV in reducing liver fibrosis of any grade, as measured by non-invasive tests, in HIV-infected people:
  * as part of a nucleoside analogue-free antiretroviral treatment regimen
  * as part of an antiretroviral treatment regimen that includes tenofovir
  Proportion of subjects with ET measurement < 5.2 kPa in the intervention group (arms 1 and 2) compared to the control group at 12 and 18 months from the start of treatment.
Efficacy of RPV in reducing liver fibrosis of any grade | 12-18 months
  Proportion of subjects with a FIB4 measurement < 1.3 in the intervention group (arms 1 and 2) compared to the control group at 12 and 18 months from the start of treatment.
Efficacy of RPV in reducing liver fibrosis of any grade | 12-18 months
  The mean reduction in the APRI measure in the intervention group (arms 1 and 2) versus the control group at 12 and 18 months after the start of treatment.
Efficacy of RPV in reducing liver fibrosis of any grade | 12-18 months
  Proportion of subjects with an APRI measure < 0.5 in the intervention group (arms 1 and 2) versus the control group at 12 and 18 months from the start of treatment.
To evaluate the efficacy of Rilpivirine (RPV) to reduce hepatic steatosis | 18 months
  The mean reduction in the percentage of liver fat, measured by magnetic resonance imaging, which measures the proton density fraction of fat (MRI-PDFF), between the beginning and the end of the study comparing the intervention group (arms 1 and 2) vs control group
To evaluate the efficacy of Rilpivirine (RPV) to reduce hepatic steatosis | 18 months
  Difference in the proportion of responders between the intervention group (arms 1 and 2) at 18 months from the start of treatment, defined as those who achieve >30% reduction in hepatic steatosis measured by MRI-PDFF
To evaluate the efficacy of Rilpivirine (RPV) to reduce hepatic steatosis | 18 months
  Proportion of subjects with hepatic steatosis measured as MRI-PDFF > 5% steatosis in the intervention group (arms 1 and 2) compared to the control group at 18 months from the start of treatment
To evaluate the efficacy of Rilpivirine (RPV) to reduce hepatic steatosis | 12-18 months
  The mean reduction of the CAP measurement in the intervention group (arms 1 and 2) compared to the control group at 12 and 18 months after the start of treatment
To evaluate the efficacy of Rilpivirine (RPV) to reduce hepatic steatosis | 12-18 months
  The mean reduction in the FLI measurement in the intervention group (arms 1 and 2) compared to the control group at 12 and 18 months after the start of treatment
To evaluate the efficacy of Rilpivirine (RPV) to reduce hepatic steatosis | 12-18 months
  The mean reduction in the HSI measure in the intervention group (arms 1 and 2) versus the control group at 12 and 18 months from the start of treatment
To evaluate the efficacy of Rilpivirine (RPV) to reduce hepatic steatosis | 12-18 months
  The mean reduction of the TyG measurement in the intervention group (arms 1 and 2) compared to the control group at 12 and 18 months after the start of treatment
To evaluate the efficacy of Rilpivirine (RPV) to reduce hepatic steatosis | 12-18 months
  Proportion of subjects with hepatic steatosis measured as CAP > 238 dB/m in the intervention group (arms 1 and 2) compared to the control group at 12 and 18 months from the start of treatment
To evaluate the efficacy of Rilpivirine (RPV) to reduce hepatic steatosis | 12-18 months
  The mean reduction in the FLI measurement in the intervention group (arms 1 and 2) compared to the control group at 12 and 18 months after the start of treatment.
To evaluate the efficacy of Rilpivirine (RPV) to reduce hepatic steatosis | 12-18 months
  Proportion of subjects with hepatic steatosis measured as HSI score > 36 in the intervention group (arms 1 and 2) versus the control group at 12 and 18 months from the start of treatment
To evaluate the efficacy of Rilpivirine (RPV) to reduce hepatic steatosis | 12-18 months
  Proportion of subjects with hepatic steatosis measured as TyG score > 8.38 in the intervention group (arms 1 and 2) compared to the control group at 12 and 18 months from the start of treatment.
To evaluate the efficacy of Rilpivirine (RPV) to decrease the insulin resistance | 12-18 months
  The mean reduction of the HOMA-IR value in the intervention group (arms 1 and 2) compared to the control group at 12 and 18 months after the start of treatment
To evaluate the efficacy of Rilpivirine (RPV) to decrease the insulin resistance | 12-18 months
  Difference in the proportion of subjects with insulin resistance, measured as HOMA-IR >2.5 in the intervention group (arms 1 and 2) versus the control group at 12 and 18 months after the start of treatment.
To evaluate the efficacy of Rilpivirine (RPV) to decrease the insulin resistance | 12-18 months
  Mean reduction in TyG (IR) measurement in the intervention group (arms 1 and 2) versus the control group at 12 and 18 months from the start of treatment.
To evaluate the efficacy of Rilpivirine (RPV) to decrease the insulin resistance | 12-18 months
  Difference in the proportion of subjects with insulin resistance measured as TyG > 4.68 in the intervention group (arms 1 and 2) compared to the control group at 12 and 18 months from the start of treatment
To evaluate the efficacy of Rilpivirine (RPV) to decrease the insulin resistance | 12-18 months
  The mean reduction in fasting blood glucose (mg/dL) in the intervention group (arms 1 and 2) versus the control group at 12 and 18 months from the start of treatment.
To evaluate the efficacy of Rilpivirine (RPV) to decrease the insulin resistance | 12-18 months
  Difference in the proportion of subjects with fasting glycemia > 100 mg/dL in the intervention group (arms 1 and 2) compared to the control group at 12 and 18 months after the start of treatment
To evaluate the efficacy of Rilpivirine (RPV) to decrease the insulin resistance | 12-18 months
  The reduction in the measurement of abdominal circumference and waist ratio/in the intervention group (arms 1 and 2) compared to the control group at 12 and 18 months after the start of treatmen
To evaluate the efficacy of Rilpivirine (RPV) to improve the lipid metabolism | 12-18 months
  The mean reduction in fasting triglycerides (mg/dL) in the intervention group (arms 1 and 2) compared to the control group at 12 and 18 months after the start of treatment.
To evaluate the efficacy of Rilpivirine (RPV) to improve the lipid metabolism | 12-18 months
  Difference in the proportion of subjects with hypertriglyceridemia (value > 150 mg/dL) in the intervention group (arms 1 and 2) compared to the control group at 12 and 18 months after the start of treatment.
To evaluate the efficacy of Rilpivirine (RPV) to improve the lipid metabolism | 12-18 months
  Mean reduction in fasting LDL cholesterol quantification (mg/dL) in the intervention group (arms 1 and 2) compared to the control group at 12 and 18 months after the start of treatment.
To evaluate the efficacy of Rilpivirine (RPV) to improve the lipid metabolism | 12-18 months
  Difference in the proportion of subjects with elevated LDL cholesterol (value > 130 mg/dL and value >100 mg/dL) in the intervention group (arms 1 and 2) compared to the control group at 12 and 18 months of start of treatment.
To evaluate the efficacy of Rilpivirine (RPV) to improve the lipid metabolism | 12-18 months
  The mean increase in fasting HDL cholesterol quantification (mg/dL) in the intervention group (arms 1 and 2) compared to the control group at 12 and 18 months after the start of treatment
To evaluate the efficacy of Rilpivirine (RPV) to improve the lipid metabolism | 12-18 months
  Difference in the proportion of subjects with elevated HDL cholesterol (value > 45 mg/dL in men and value > 50 mg/dL in women) in the intervention group (arms 1 and 2) compared to the control group at 12 and 18 months from the start of treatment
To evaluate the efficacy of Rilpivirine (RPV) to improve the lipid metabolism | 12-18 months
  The mean reduction in fasting non-LDL cholesterol quantification (mg/dL) in the intervention group (arms 1 and 2) compared to the control group at 12 and 18 months after the start of treatment.
To evaluate the efficacy of Rilpivirine (RPV) to improve the lipid metabolism | 12-18 months
  Difference in the proportion of subjects with elevated non-LDL cholesterol (value > 160 mg/dL) in the intervention group (arms 1 and 2) compared to the control group at 12 and 18 months after the start of treatment
To evaluate the efficacy of Rilpivirine (RPV) to decrease the liver inflammation | 12-18 months
  The mean change in ALT value (IU/mL) in the intervention group (arms 1 and 2) vs. the control group at 12 and 18 months from baseline
To evaluate the efficacy of Rilpivirine (RPV) to decrease the liver inflammation | 12-18 months
  The mean change in AST value (IU/mL) in the intervention group (arms 1 and 2) versus the control group at 12 and 18 months from the baseline visit
To evaluate the efficacy of Rilpivirine (RPV) to decrease the liver inflammation. | 12-18 months
  The change of the gene expression value of: IL1-beta, IL6, IL10, MCP1, PAI-1, TGF-alpha, TNF-alpha in PBMCs in the intervention group (arms 1 and 2) compared to the control group at 12 and 18 months compared to the baseline visit.
Efficacy of RPV to reduce hepatic steatosis/fibrosis. | 18 months
  To assess the efficacy of RPV as part of the antiretroviral treatment regimen in HIV-infected individuals to reduce hepatic steatosis/fibrosis based on the presence of PNPLA3 and MBOAT7-TMC4 genetic polymorphisms.
To characterise the effects of RPV on the expression of inflammatory and fibrogenic markers in peripheral blood mononuclear cells | 18 months
  . Analyse the gene expression of inflammatory and fibrogenic markers in peripheral blood polymorphonuclear cells by RT-PCR: IL1-gamma, IL6, IL10, MCP1, P AI-1, TGF-beta, TNF-alpha.
To characterise the effects of RPV on the expression of inflammatory and fibrogenic markers in peripheral blood mononuclear cells | 18 months
  . Measurement of ALT, AST and GGT in plasma as markers of inflammation.
Efficacy of RPV to reduce the progression to steatohepatitis | 18 months
  In previous studies it has shown that PNPLA3, TM6SF2, and MBOAT7-TMC4 polymorphisms are associated with elevated ALT levels and histologic parameters of nonalcoholic steatohepatitis and fibrosis severity.
  On the baseline visit will be collected biological samples for genetuic study. A 3 ml blood sample will be drawn into an EDTA tube at baseline visit for determination of PNPLA3 (C, G alleles) and MBOAT7-TMC4 (G, A alleles) genetic polymorphisms.

CONTACTS AND LOCATIONS:
Locations (4):
- Spain (4):
  - Hospital Universitario Gregorio Marañon, Madrid
  - Hospital universitario Infanta Leonor, Madrid
  - Hospital Universitario Infanta Sofía, Madrid
  - Hospital Universitario La Paz, Madrid